CLINICAL TRIAL: NCT00562146
Title: Rate of Postpyloric Migration of Spiral Nasojejunal Tubes in Brain Injured Patients
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Jian-Xin Zhou, ICU, Beijing Tiantan Hospital, Capital Medical University
Other Study IDs: BJTTH-ICU-07-011; BJTTH-ICU-07-011
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Acute Brain Injury
Keywords: nutrition; enteral access
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Successful progression of spiral tube to duodenum within 3 days
  Interventions: Procedure: placement of spiral nasojejunal tube
- 2: Failure of progression to duodenum within 3 days
  Interventions: Procedure: placement of spiral nasojejunal tube

INTERVENTIONS:
Procedure: placement of spiral nasojejunal tube — spiral nasojejunal tube will be placed after enrollment of the patients

SUMMARY:
The success rate of unguided nasojejunal feeding tube insertion will be determined in acute brain injured patients. Factors influencing tube self-progression will be evaluated.

DETAILED DESCRIPTION:
Nutrition support is important in brain injured patients. Several studies have shown that small bowel feeding compared with gastric feeding may be associated with a reduction in pneumonia in critically ill patients. The Canadian Clinical Practice Guidelines recommended that small bowel feedings should be considered for patients at high risk for intolerance to enteral nutrition.

There are several methods to place postpyloric tube, but there is a high success rate with endoscopic or radiological assistance. However, they are time consuming procedures, which is of limited availability at bedside and requires trained staff.

Nasojejunal tube with spiral end (Flocare Bengmark NJ tube) has been used for bedside placement for 10 years. But only limited data are available for success rate, especially in brain injured patients. The aim of this study is to access the success rate and influencing factors of spiral end nasojejunal tube in such a population.

ELIGIBILITY:
Inclusion Criteria:

* Acute brain injured patients admitted to Neuro-ICU

Exclusion Criteria:

* Patients' stay in ICU shorter than 3 days
* Patients with contraindication to naso-feeding tube placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute brain injured patients admitted to Neuro-ICU will be consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Study Chair — ICU, Beijing Tiantan Hospital, Capital Medical University
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China